CLINICAL TRIAL: NCT05816655
Title: Comparison of Clinical Efficacy Between Letrozole + Ribociclib and Fulvestrant + Letrozole + Ribociclib in Hormone Receptor Positive, HER2 Negative Metastatic Breast Cancer - a Randomized, Phase 2 Study
Brief Title: Comparison of Clinical Efficacy Between Letrozole + Ribociclib and Fulvestrant + Letrozole + Ribociclib in Hormone Receptor Positive, HER2 Negative Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Park, In Hae, Principal investigator, Clinical professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCSG BR22-20
Record Dates: First submitted 2023-03-22; First posted 2023-04-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fulvestrant arm (Experimental): fulvestrant + AI + ribociclib
  Interventions: Drug: Fulvestrant plus AI plus ribociclib
- Control arm (Active Comparator): AI + ribociclib
  Interventions: Drug: AI plus ribociclib

INTERVENTIONS:
Drug: Fulvestrant plus AI plus ribociclib — Fulvestrant + AI + ribociclib +/- GnRH agonist
  Arms: Fulvestrant arm
Drug: AI plus ribociclib — AI + ribociclib +/- GnRH agonist
  Arms: Control arm

SUMMARY:
Aromatase inhibitor (AI) + CDK4/6 inhibitor is settled down as the standard first line therapy for HR+/HER2- metastatic breast cancer and all three CDk4/6 inhibitors, palbociclib, ribociclib, and abemaciclib are currently available for same indications. However, there is no effective treatment strategy for patients who have progressed on AI+CDK4/6 inhibitor. In particular, the clinical efficacies of subsequent hormone therapy are lowered when ESR1 mutations, one of mechanisms of AI resistance occur. In the PADA-1 trial, when ESR1 mutations in ctDNA were detected in patients treated with AI+CDK4/6 inhibitor, AI was switched to fulvestrant even if disease progression was not confirmed clinically. As a result, the median PFS was prolonged by about 8 months in this switching group compared to the group in which AI was continued. The results of this study suggested that delaying the occurrence of ESR1 mutations and early response to them are necessary to increase the effectiveness of hormone therapy.

In SWOG S0226 study, fulvestrant + AI combination showed significant benefits in PFS and OS compared to AI monotherapy as the first line therapy. Based on these results, the NCCN guideline suggests fulvestrant + AI combination as one of the first line hormone therapy options. However, the clinical effect of AI + fulvestrant + CDK4/6 inhibitor has not been investigated yet. Therefore, the investigators are planning to compare the clinical efficacy of AI+ fulvestrant + CDK4/6 inhibitor and AI+CDK4/6 inhibitor, and to investigate if a triple combination regimen can delay the emergence of ESR1 mutations and modulate occurred ESR1 mutations.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 19 years of age
* Histologically confirmed unresectable, locally advanced or metastatic invasive breast cancer with hormone receptor positive/HER2 negative
* No previous history of systemic endocrine or chemotherapy for metastatic, advanced breast cancer.
* If the patient has received AI as adjuvant endocrine therapy, the treatment free interval (TFI) should be more than 12 months after the end of adjuvant endocrine therapy. If the patient has received tamoxifen for adjuvant endocrine therapy, TFI less than 12 months will be allowed.
* ECOG PS 0-2
* Patients should have measurable or evaluable lesion based on RECIST version 1.1
* Patients should have adequate organ function:

  * ANC (absolute neutrophil count) ≥ 1.5 × 109/L
  * Platelet ≥ 100 × 109/L
  * Serum Hb ≥ 9.0 g/dL
  * INR ≤1.5
  * Serum creatinine ≤ 1.5 X ULN
  * ALT & ALT <2.5 X ULN, if patients have hepatic metastasis, ALT & ALT <5.0 X ULN is allowed
  * Total serum bilirubin <1.5 X ULN, if patients have hepatic metastasis, Total serum bilirubin <3.0 X ULN is allowed.
* In the case of childbearing potential, patients who can adhere to appropriate contraception during the study period and for at least 6 months after the end of study treatment.
* Patients who understand the contents of the clinical trial and are cooperative with the process of the clinical trial.

Exclusion Criteria:

* Patients with a history of previous treatment with a CDK4/6 inhibitor or other systemic treatment for advanced/metastatic breast cancer
* Patients who have received prior treatment with fulvestrant and any investigational ER-directed therapy including SERDs (selective estrogen receptor degrader)
* Patients who have disease recurrence on aromatase inhibitor treatment as adjuvant endocrine therapy
* Patients who have symptomatic or untreated central nervous system metastasis
* Patients who have a history of cardiovascular disease or heart failure as following conditions; within at least 6 months of myocardial infarction, unstable angina, or uncontrolled arrhythmia.
* Patients having visceral crisis which needs rapid tumor reduction
* Patients who have a history of any other cancer (except nonmelanoma skin cancer, carcinoma in-situ of the cervix, well-differentiated thyroid cancer)
* Patients unable to cooperate with periodic blood samples collection
* Patients who have active HBV, HCV infection, immune-suppressive disease, or HIV infection. In case of chronic HBV infection, HBV DNA should be negative. Patients with complete remission of HCV infection are allowed.
* Pregnant or breast-feeding women
* Patients who are considered to be unsuitable for this trial by investigators.

Ages: 19 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
24 month- progression free survival rate | the time from randomization until documented disease progression or death from any cause, whichever occurs first, assessed up to 24 months.
  To compare 24 month- progression free survival rate (PFS rate) of letrozole + ribociclib + fulvestrant to letrozole + ribociclib for HR+/HER2- metastatic breast cancer (MBC) as the 1st line endocrine therapy

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Korea university Guro hospital, Seoul
  - St Mary Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided